CLINICAL TRIAL: NCT04920318
Title: Enhancing Language Function in Primary Progressive Aphasia (PPA) With Transcranial Direct Current Stimulation (tDCS)
Brief Title: Enhancing Language Function in Primary Progressive Aphasia
Acronym: PPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2103570362
Record Dates: First submitted 2021-06-01; First posted 2021-06-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Primary Progressive Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Transcranial Direct Current Stimulation; Language Therapy

STUDY DESIGN:
Intervention Model Description: individuals diagnosed with Alzheimer's Disease Primary Progressive Aphasia (AD-PPA) (~50-80 years old) will be randomized to receive active tDCS+language treatment or sham (fake tDCS)+language treatment in a cross-over design.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subject codes will be used for blinding of the participants, care-providers, and speech-language therapist administering the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active TDCS (Experimental): During intervention excitatory/anodal tDCS will be administered alongside speech-language therapy 5 days a week for 2 weeks. The exact location of the stimulation and electrode configuration will be targeted individually based on the optimal site identified in fMRI. TDCS will be administered with NeurConn1 Channel DC- Stimulator Plus (neuroCare Group, München, Germany) according to established guidelines and procedures. The active tDCS will be delivered for 20 minutes using sponge electrodes with a 30-s ramp-up and ramp-down period
  Interventions: Combination Product: tDCS + language therapy
- sham TDCS (Sham Comparator): The sham will be administered alongside speech-language therapy 5 days a week for 2 weeks. For sham, stimulation will be ramped up and then down to 0 milliamperes (mA) in the first minute of stimulation. The sham parameters were chosen based on previous reports that the perceived sensations on the skin, such as tingling, fade out in the first 30 s of tDCS
  Interventions: Combination Product: sham TDCS + language therapy

INTERVENTIONS:
Combination Product: tDCS + language therapy — In this study fMRI-guided noninvasive neuromodulation will be applied, called Transcranial Direct Current Stimulation (tDCS) to the frontal and parietal brain regions that show reduced activation but still are structurally intact. TDCS will be paired with personalized speech-language therapy to enhance language functions.
  Other Names: active tDCS; transcranial direct current simulation (tDCS)
  Arms: active TDCS
Combination Product: sham TDCS + language therapy — sham control will be applied with language therapy to the same regions as active TDCS.
  Other Names: sham transcranial direct current simulation (tDCS)
  Arms: sham TDCS

SUMMARY:
This study's goal is to use non-invasive brain stimulation (NBS) techniques to treat language impairment associated with Primary Progressive Aphasia (PPA). The purpose of this study is to combine behavioral language intervention with individualized noninvasive brain stimulation techniques, called transcranial direct current stimulation (tDCS) to help the brain reorganize around damage and improve language functions.

DETAILED DESCRIPTION:
Primary Progressive Aphasia (PPA) is a neurodegenerative disorder that selectively affects language comprehension and/or production, with initial preservation of other cognitive domains. As tDCS has not been extensively studied in PPA, the investigators will measure both short- and long-term effects of stimulation in patients with this neurodegenerative disorder that affects specific language regions. Previous research suggests that neurostimulation with tDCS can safely induce changes in neural plasticity that can lead to long-term restoration of synaptic function. Thus, individually targeted stimulation to structurally preserved but dysfunctional regions may be able to produce behavioral improvements in primary progressive aphasia (PPA).

TDCS is a method of stimulating the brain that does not require any sedation or surgery. TDCS is a technique that sends a weak electrical current through the scalp to stimulate the brain areas below. The information gained from this research study will aid in the development of therapies to improve language in people with neurological conditions that affect language use.

TDCS will be applied over the activated area identified with the functional magnetic resonance imaging (fMRI) fMRI-localizer task. This approach will allow for individually optimized tDCS electrode placement. It will also account for potential inter-participant variability in the brain atrophy and language organization

Summary of study sequence and procedures:

Week 1: Baseline screening, language testing, one event-related brain potential (EEG-ERP) session Weeks 2: fMRI session to determine most effective treatment Weeks 3-4: tDCS with Language Treatment Part 1 Weeks 5 and 6: rest-period, post-treatment assessment Weeks 7 to 8: TDCS with Language Treatment Part 2 Weeks 9 and 10: rest period, post-treatment assessment 2-month follow-up, language assessment, one MRI scan, one EEG-ERP session

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PPA by neurologist or speech-language pathologist
* speech-language deficit arising from PPA
* native speaker of English Language or equivalent
* adequate vision (normal or corrected to normal)
* adequate hearing

Exclusion Criteria:

* meeting (Diagnostic and Statistical Manual) DSM-IV criteria for Axis I mood, anxiety, psychotic or substance abuse disorders.
* highly magnetizable metallic implants, including certain dental work
* neurological disorders besides the ones of interest for the study (e.g., epilepsy)
* Multiple Sclerosis
* Parkinson's Disease
* contraindications for MRI
* pacemakers
* metallic cardiac pumps
* valves
* magnetic materials such as surgical clips, implanted electronic perfusion pumps, or any other condition that would preclude proximity to a strong magnetic field.
* clinically significant claustrophobia
* severe systemic disease (e.g., renal failure)
* poor health
* pregnancy
* epileptic activity in the past 12 months
* family history of epilepsy or other seizure disorders
* brain surgery in the past
* metallic skull plates or implants
* skin lesions or skull damage
* excessive use of alcohol or drugs
* premorbid psychiatric disease affecting communication
* severe non-linguistic cognitive disturbances impeding language therapy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline scores on the Arizona Phonological Battery | through study completion, an average of 1 year
  Mean change from baseline scores on the Arizona Phonological Battery: Minimum score = 0; maximum = 100%; higher scores indicate better outcome
Mean change from baseline scores on the naming task | through study completion, an average of 1 year
  Mean change from baseline scores on the Boston Naming Test: Min score = 0; Max = 60; higher scores indicate better outcome
Mean change from baseline scores on the language probe task before and after each session | through study completion, an average of 1 year
  change on on the probe task from before the session; Min =0; Max = 100%; higher scores indicate better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Aneta Kielar, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No